CLINICAL TRIAL: NCT01261741
Title: Prospective, Randomized, Double-blind, Placebo-controlled, Multi-center Study to Investigate the Efficacy and Safety of 10mg Memantine in the Treatment of Memory, Concentration or Attention Problems in the Absence of Dementia
Brief Title: Investigation of Memantine in the Treatment of Memory, Concentration or Attention Problems
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MRZ 90001-2267 / 1; 2010-020737-50 (EudraCT Number)
Record Dates: First submitted 2010-12-15; First posted 2010-12-16 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Memory Disorder; Retention Disorder, Cognitive; Subjective Cognitive Impairment; Memory, Concentration or Attention Problems
MeSH Terms: conditions — Memory Disorders | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Memantine (Experimental)
  Interventions: Drug: Memantine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Memantine — Each subject will receive memantine 10mg tablets once daily
  Arms: Memantine
Drug: Placebo — Each subject will receive matching placebo tablets once daily
  Arms: Placebo

SUMMARY:
In this study, memantine will be tested in a new indication: in the treatment of subjective memory, concentration, or attention problems (subjective cognitive impairment) in the absence of dementia.

ELIGIBILITY:
Inclusion Criteria:

* Subjective worsening of memory, concentration or attention problems for longer than 6 months
* Subject can confirm that a relative or friend has noticed the memory, concentration or attention problems of the subject
* Experience of the memory, concentration or attention problems at least four times per week

Exclusion Criteria:

* Significant neurological disease or major psychiatric disorder (e.g. diagnosis of psychosis or dementia)
* Significant systemic illness, such as cancer, heart or kidney failure, uncontrolled diabetes
* History of stroke or seizure, or myocardial infarction within the last year (e.g. by inclusion questionnaire, physician interview)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2010-11; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
"Patient Global Impression of Change" (PGI-C) at visit 4 | 12 weeks
  It is the statistical comparison between the placebo group and the memantine group.The group comparison will be performed by the use of an analysis of covariance (ANCOVA) model.

SECONDARY OUTCOMES:
Change from baseline to visit 3 and 5 of Patient Global Impression of Change (PGI-C) | 16 weeks
Change from baseline to visit 4 in "Everyday Cognition 39" (ECog 39) total score | 12 weeks
Change from baseline to visit 4 in "Hospital Anxiety and Depression Scale" (HADS) Score | 12 weeks
Change from baseline to visit 3, 4, 5 of "Computer-based Neuropsychological Test Battery (C-NTB) by CogState Ltd. | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Merz Medical Expert, Study Director — Merz Pharmaceuticals GmbH
Locations (14):
- Germany (11):
  - Universitätsklinikum der RWTH Aachen, Aachen
  - Praxis Dr. Heidenreich, Böblingen
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Praxis Dr. Albrecht, Ellwangen
  - Praxis Dr. Reifschneider, Erbach im Odenwald
  - Klinische Forschung Hannover-Mitte, Hanover
  - ZSL Zentrum für medizinische Studien in Leipzig, Leipzig
  - Klinische Forschung Berlin-Mitte, Mitte
  - Praxis Dr. Pauls, München
  - Praxis Dr. Kühn, Oranienburg
  - Praxis Dr. Krause, Wolfratshausen
- United Kingdom (3):
  - Royal United Hospital, Bath
  - Community Pharmacology Services (CPS), Glasgow
  - Moorgreen Hospital, West End, Southampton

REFERENCES:
- [Result] Schulz JB, Acker C, Seitzinger A, Pulte I. Randomized, double-blind, placebo-controlled, multicentre study to investigate memantine in the treatment of memory, concentration, and attention problems (subjective cognitive impairment). Journal of the Neurological Sciences 333 Suppl.1: e332, 2013. doi:10.1016/j.jns.2013.07.1232